CLINICAL TRIAL: NCT07378020
Title: Comparative Study Between Densah Burs Versus Osteotome Preparation in Implant Stability Placed in Areas of Low Bone Density.
Brief Title: Comparing Between Densah Burs Versus Osteotome in Low Bone Density Areas.
Acronym: osseo-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Mohamed Mahmoud, Principal Investigator, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUE.REC (25)/7-2023
Record Dates: First submitted 2026-01-18; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Low Bone Density
Keywords: Osseodensification
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant
Masking Description: A randomization sequence was generated using a web-based service (Randomization.com) employing block randomization. To ensure allocation concealment, a research coordinator (who was not involved in the clinical procedures) prepared sequentially numbered, opaque, sealed envelopes corresponding to the total number of implants required for the study. At the time of surgery, a research colleague opened the next sequential envelope for each implant site to determine the group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Drilling (Active Comparator): Implant sites in this arm will undergo osteotomy preparation using standard conventional drilling sequences according to the implant manufacturer's recommendations prior to implant placement
  Interventions: Procedure: Conventional Osteotomy
- Densah Bur (Osseodensification) (Experimental): Implant sites in this arm will undergo osteotomy preparation using the osseodensification technique with Densah burs (Versah) running in a counter-clockwise direction (densifying mode) prior to implant placement.
  Interventions: Procedure: Densah Bur drilling
- osteotome (Experimental): Implant sites in this arm will undergo osteotomy preparation using summers osteotome technique for lateral bone condensation and expansion prior to implant placement
  Interventions: Procedure: osteotome bone condensation

INTERVENTIONS:
Procedure: Conventional Osteotomy — The implant site will be prepared using a standard sequence of drills (subtractive osteotomy) according to the implant manufacturer's instructions. Drilling will be performed with profuse irrigation at speed between 800-1200 rpm to remove bone and prepare the osteotomy site to the final diameter before implant insertion
  Other Names: Subtractive Drilling; Standard Drilling
  Arms: Conventional Drilling
Procedure: Densah Bur drilling — after using the pilot drill in a clockwise direction to drill to the desired depth according to the planned implant length The implant site will be prepared using Densah burs (Versah). the motor is adjusted to rotate in a counter-clockwise direction (densifying mode) at 800-1200 rpm with profuse irrigation. This technique expands the osteotomy site by compacting bone at the periphery rather than removing it, aiming to enhance bone density around the implant then the implant is inserted after reaching the desired diameter according to densah bur soft bone drilling protocol
  Other Names: Osseodensification; Non-subtractive Drilling
  Arms: Densah Bur (Osseodensification)
Procedure: osteotome bone condensation — osteotomy was prepared using (Xive BoneCondensers by dentsply sirona GERMANY) starting from the pilot drill of 1.7mm in diameter to penetrate the cortical bone and gain access. Then instrumentation was done in the following sequence: 2.0mm, 3.0mm, and 3.4mm according to the planned implant diameter. The osteotome was inserted manually and rotated while being pressed towards the apical part of osteotomy till it reaches the full working depth. Once the desired depth was reached, and before moving to the next instrument we wait 1 min for the osteotome to compress and compact the spongy bone. After the implant bed had been prepared, we inserted the implant immediately to avoid any dimensional changes in the site of osteotomy.
  Other Names: Manual Bone Condensation; Osteotome Expansion
  Arms: osteotome

SUMMARY:
The objective of this study is to compare the primary stability of implant sites prepared using conventional drilling, osseodensification (Densah bur), and osteotome preparation techniques, and to evaluate the influence of these methods on implant success rates in areas of low bone density.

DETAILED DESCRIPTION:
in different conditions implants that lack primary stability is subjected to excessive micromotion that can lead to implant failure. This usually happens when dental implants pass the critical limit of micro-motion. Passing this critical limit can interfere with Osseo-integration and cause fibrous encapsulation of dental implant .

Implant Failure usually occurs in completely edentulous maxillae especially in the posterior area where bone quality is compromised.

Clinicians usually refer implants success rates to the difference in bone quality between mandible and maxilla. Higher failure rates seem to be associated with poor bone quality.

Primary stability is affected by several factors including Bone Quantity and quality, the Implant macro- and micro- design, and the used osteotomy technique.

Osteotomies are usually created using conventional drills, although the implant diameter must be slightly larger than the final drill to ensure primary stability However, this conventional drilling technique might be insufficient to provide the primary stability required for Osseo-integration in areas of low bone quality. Several site preparation techniques have been introduced to enhance primary stability in soft bone. Some clinicians used under-sized drilling however the efficiency of this technique is conditioned by decreasing osteotomy diameter by 10% of implant diameter.

Another method introduced by Dr. Robert Summer. This method uses bone condensers to densify bone through the condensation and expansion of spongy bone as it squeezes bone trabeculae laterally against the wall of implant bed at the site of osteotomy increasing the bone density and conserving osseous tissue around implants.

Recently Osseodensification (OD) was introduced as a novel implant site preparation technique that uses specially designed drills with large negative rake angles. When the drills are operated in a counterclockwise direction it acts as a non-cutting drill which is used to expand and compact bone against the osteotomy walls. This non-subtractive approach aims to increase the primary stability of the dental implants inserted into low-density bone compared with conventional drilling techniques. The drills also can be used as a cutting drill when operated in a clockwise direction according to the operator's need. This type of drill can improve bone density leading to improved implant primary stability, giving these drills the ability to cut and densify without the need for additional tools.

Ossoe-densification technique showed greater insertion torques, bone-to implant contact, and bone area fraction occupancy when compared to standard Drilling technique.

this study is comparing between the three different drilling techniques (conventional, osseo-densification, osteotome bone compaction) in enhancing insertion torque and isq values in posterior maxillary area.

the study also compare between the effect of these techniques on marginal bone loss with follow up 6 month after loading using cbct

ELIGIBILITY:
Inclusion Criteria:

* Patients with low bone density (D3), (D4) Missing maxillary posterior teeth
* edentulous ridge should be 8 mm or more of bone height and bone width ≥ 7mm with adequate inter-occlusal space of at least 8mm,
* Patients with good oral hygiene or willing to improve their oral hygiene.

Exclusion Criteria:

* Patients with uncontrolled medical conditions that affect Osseo-integration.
* Patients receiving medications that contraindicate osteotomy.
* Heavy smokers.
* History of receiving irradiation in the head and neck region.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2025-01-05 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
primary stability using Insertion Torque Value. | day of surgery
  Evaluation of implant stability was done by measuring Insertion torque. Using the surgical contra-angled hand piece the initial torque value was set to10Ncm then increased sequentially by 5Ncm according to the torque required to place the implant at the desired depth. The final torque value used to drive the implant to its position was recorded as the peak insertion torque
Primary Implant Stability measured through Resonance Frequency Analysis (RFA) | the day of surgery
  Implant stability will be measured using Resonance Frequency Analysis (RFA) via an Osstell device. The values are recorded as Implant Stability Quotient (ISQ) on a scale from 1 to 100, where higher scores indicate greater stability

SECONDARY OUTCOMES:
Secondary Implant Stability using radio frequency analysis (RFA) | readings were taken 3 months post operative and 6 months after loading.
  Implant stability measured using Resonance Frequency Analysis (RFA) via Osstell. Values recorded as ISQ (1-100) to evaluate osseointegration. where higher scores indicates higher stability
Marginal Bone Loss (MBL) | cbct was done at implant placement and 3 months post operative and 6 months after loading.
  Radiographic evaluation of crestal bone changes measured using cone beam CT. The difference in bone level between baseline and follow-up will be calculated in millimeters.

CONTACTS AND LOCATIONS:
Overall Officials: dr lobna abdelaziz aly, PhD, Study Director — Future University in Egypt
Locations (1):
- Oral and Maxillofacial Department Future Dental Hospital, Cairo, Fifth Settlement, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elsheikh HA, Gadallah AT, Kandil I. Impact of Three Different Surgical Drilling Protocols on Early Loaded Single Implant in Posterior Maxilla: A 3-year Follow-up. J Contemp Dent Pract. 2022 Aug 1;23(8):819-827.
- [Background] Evrenk O, et al. Evaluation of implant primary stability using different drilling protocols: an in vitro study. BMC Oral Health. 2025 Aug 9. doi: 10.1186/s12903-025-06661-4.
- [Background] Huwais S, Meyer EG. A Novel Osseous Densification Approach in Implant Osteotomy Preparation to Increase Biomechanical Primary Stability, Bone Mineral Density, and Bone-to-Implant Contact. Int J Oral Maxillofac Implants. 2017 Jan/Feb;32(1):27-36.
- [Background] Summers RB. A new concept in maxillary implant surgery: the osteotome technique. Compend Contin Educ Dent. 1994 Feb;15(2):152, 154-6, 158 passim.